CLINICAL TRIAL: NCT04641897
Title: Impact of Decreasing Respiratory Rate, While Tolerating Moderate Hypercapnia, on Lung Injury Markers in Patients with Acute Respiratory Distress Syndrome
Brief Title: Impact of Decreasing Respiratory Rate on Lung Injury Biomarkers in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 180813016; 1191315 (Other Grant/Funding Number: Fondecyt)
Record Dates: First submitted 2020-10-09; First posted 2020-11-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2020-11

CONDITIONS: Acute Respiratory Distress Syndrome; Respiration, Artificial; Ventilator-Induced Lung Injury
Keywords: Respiratory rate; Mechanical ventilation; ARDS; Ventilator induced lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Other): Sequence A: Low RR for 12 hours - High RR for 12 hours
  Interventions: Procedure: Respiratory rate modification
- Sequence B (Other): Sequence B: High RR for 12 hours - Low RR for 12 hours.
  Interventions: Procedure: Respiratory rate modification

INTERVENTIONS:
Procedure: Respiratory rate modification — During the Low RR and High RR periods, respiratory rate will be set depending on baseline ABG and according a nomogram so as to have an approximate difference of 10 points between groups, while maintining PaCO2 and pH values within safety limits (pH 7.20 to 7.45, and PaCO2 35 to 60 mmHg).
  Once defined the target respiratory rate, this will be decreased or increased in 4 points each 30 to 45 min, and ABG repeated at 2 hours. At this time, changes will be made to keep PaCO2 and pH values within safety limits, and ABG repeated at 6 and finally 12 hours.
  During the whole period, inspiratory to expiratory ratio will be maintained constant, and only changed to keep inspiratory time above 0.6 seconds (usually at high resp rate).

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a form of acute lung injury of inflammatory origin, which represents a public health problem worldwide due to its prevalence, and its high mortality rate, close to 40%. Mechanical ventilation is a fundamental therapy to improve gas exchange, however, it can also induce further lung injury, a phenomenon known as ventilator induced lung injury (VILI). The limitation of tidal volume is the strategy that has shown the greatest decrease in mortality and is the cornerstone of protective ventilation. However, the respiratory rate, a fundamental parameter in the programming of the mechanical ventilator, has not been evaluated in most of the main clinical studies to date. Moreover, the natural clinical response to the use of a low tidal volume strategy is the increase in respiratory rate, which may harm the lung as it increases the energy applied to the lung parenchyma. The investigators hypothesize that the use of a lower respiratory rate, tolerating moderate hypercapnia, is associated with less VILI, measured by the release of proinflammatory mediators at the systemic level (biotrauma), compared to a conventional higher respiratory rate strategy in patients with moderate to severe ARDS. This effect is mediated by lower energy applied to the pulmonary parenchyma. To confirm this hypothesis the investigators propose a prospective cross-over clinical trial in 30 adult patients with ARDS in its acute phase, which will be randomized to two sequences of ventilation. Each period will last 12 hours, and respiratory rate (RR) will be set according to PaCO2 goal: 1) Low RR, PaCO2 60-70 mmHg; and 2) High RR, PaCO2 35-40 mmHg.

Protective ventilation will be applied according to ICU standards under continuous sedation and neuromuscular blockade. Invasive systemic arterial pressure and extravascular lung water will be monitored through an arterial catheter (PICCO® system), and airway and esophageal pressures and hemodynamics continuously measured throughout the protocol. The main outcome will be Interleukin-6 in plasma. At baseline and at the end of each period blood samples will be taken for analysis, and electrical impedance tomography (EIT) and transthoracic echocardiography will be registered. After the protocol, patients will continue their management according to ICU standards.

ELIGIBILITY:
Inclusion Criteria:

Patients intubated and under mechanical ventilation with acute respiratory distress syndrome less than 48 hours

1. Acute onset (less than 1 week)
2. Chest-X-ray: bilateral infiltrates
3. Absence of heart failure or hydrostatic pulmonary edema
4. Oxygenation disorder: PaO2/FiO2 ratio <200, with PEEP ≥5 cmH2O

Exclusion Criteria:

* Age <18 years
* Previous chronic respiratory disease (chronic obstructive lung disease, asthma, intersticial lung disease, pulmonary fibrosis, chronic bronchiectasis)
* Hypercapnic respiratory failure, defined as PaCO2 >60 mmHg or pH<7.25 despite a RR >30.
* Concomitant severe metabolic acidosis: pH<7.20
* Catastrophic respiratory failure, defined as PaO2/FiO2 ratio <80, despite optimization of ventilatory parameters, or need for ECMO.
* Contraindication to hypercapnia, such as intracranial hypertension or acute coronary syndrome
* Use of vasoconstrictor drugs in increasing doses in the last 2 hours (≥0.5 μg/kg/min of noradrenaline) or average blood pressure <65mmHg
* Pneumothorax or subcutaneous emphysema, not drained.
* Pregnancy
* Presence of mental or intellectual disability prior to hospitalization
* Early limitation of therapeutic effort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in IL-6 | baseline, 12 and 24 hours
  levels of IL-6 in plasma

SECONDARY OUTCOMES:
Changes in transpulmonary driving pressures | Baseline, 12 and 24 hours
Changes in Auto PEEP | Baseline, 12 and 24 hours
Changes in mean airway pressure | Baseline, 12 and 24 hours
Changes in level of energy applied to the lungs | Baseline, 12 and 24 hours
Changes in arterials blood gases | Baseline, 12 and 24 hours
Changes overtime in distribution of ventilation | Baseline, 6,12, 24 hours
  Distribution of ventilation as assessed by Electrical impedance tomography
Changes in cardiac function and pulmonary edema | Baseline, 12 and 24 hours
  measured by PICCO®.
Changes pulmonary edema | Baseline, 12 and 24 hours
  measured by PICCO®.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad Catolica, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damiani LF, Basoalto R, Oviedo V, Alegria L, Soto D, Bachmann MC, Jalil Y, Santis C, Carpio D, Ulloa R, Valenzuela D, Vera M, Schultz MJ, Retamal J, Bruhn A, Bugedo G. Effect of decreasing respiratory rate on the mechanical power of ventilation and lung injury biomarkers: a randomized cross-over clinical study in COVID-19 ARDS patients. Intensive Care Med Exp. 2025 Jul 9;13(1):69. doi: 10.1186/s40635-025-00782-4. PMID 40632387